CLINICAL TRIAL: NCT01404741
Title: Comparison Between 5-azacytidine Treatment and 5-azacytidine Followed by Allogeneic Stem Cell Transplantation in Elderly Patients With Advanced MDS According to Donor Availability
Brief Title: 5-azacytidine Treatment Versus 5-azacytidine Followed by Allogeneic Stem Cell Transplantation in Elderly Patients With Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: VidazaAlloStudy
Record Dates: First submitted 2011-06-30; First posted 2011-07-28 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia
Keywords: MDS; CMML; allogeneic stem cell transplantation; 5-azacytidine
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-azacytidine treatment until progress (Active Comparator): 5-azacytidine until progress
  Interventions: Procedure: 5-azacytidine until progress
- allogeneic stem cell transplantation (Experimental): after 4 cycles 5-azacytidine and if donor available: allogeneic stem cell transplantation after reduced intensity conditioning
  Interventions: Procedure: allogeneic stem cell transplantation

INTERVENTIONS:
Procedure: allogeneic stem cell transplantation — donor available, after 4 cycles 5-azacytidine allogeneic stem cell transplantation after reduced conditioning
  Arms: allogeneic stem cell transplantation
Procedure: 5-azacytidine until progress — if no donor available 5-azacytidine until progress or toxicities
  Arms: 5-azacytidine treatment until progress

SUMMARY:
5-azacytidine treatment prolongs survival in patients with myelodysplastic syndrome (MDS), but does not cure the disease. Allogeneic stem cell transplantation is a curative treatment option but is associated with a high risk treatment-related morbidity and mortality. In the current trial allogeneic stem cell transplantation will be compared to 5-azacytidine only treatment according to donor availability in elderly patients with MDS (55-70 years).

DETAILED DESCRIPTION:
5-azacytidine treatment prolongs survival in patients with myelodysplastic syndrome (MDS), but does not cure the disease. Allogeneic stem cell transplantation is a curative treatment option but is associated with a high risk treatment-related morbidity and mortality. Dose-reduced conditioning prior transplantation allows also treatment of elderly patients with MDS. In the current trial allogeneic stem cell transplantation will be compared to 5-azacytidine only treatment according to donor availability in elderly patients with MDS (55-70 years).

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven de novo or therapy-related MDS / CMML (WBC <13 GPT/l)according to FAB and risk profile according to IPSS: intermediate II- risk or high-risk or intermediate I with high-risk cytogenetic (according to IPSS, taking into account that IPSS, however, was not validated for t- MDS), patients with secondary AML (according to WHO) and blasts ≤ 30 % (= RAEB-t according to FAB)
* Previously untreated or maximal 1 cycle of 5-azacytidine (Vidaza®)
* Male or Female; Age 55 - 70 years
* Understand and voluntarily sign an informed consent form
* ECOG performance status of ≤ 2 at study entry
* Adequate renal and liver function: creatinine and bilirubin < 3 x the upper limit of normal
* Sufficient cardiac function (ejection fraction > 30 %)

Exclusion Criteria:

* Blasts > 30 % in bone marrow at time of diagnosis
* Central nervous involvement
* Severe irreversible renal, hepatic, pulmonary or cardiac disease, such as
* Total bilirubin, SGPT or SGOT ≥ 3 times upper the normal level
* Left ventricular ejection fraction < 30 %
* Creatinine clearance < 30 ml/min
* DLCO < 35 % and/or receiving supplementary continuous oxygen
* Pregnant or breastfeeding female subject
* Patients with a life-expectancy of less than six months because of another debilitating disease
* Serious psychiatric or psychological disorders
* Uncontrolled invasive fungal infection at time of registration
* Known positive for HIV or acute infectious hepatitis, type A, B or C
* Participation in another study with ongoing use of unlicensed investigational product from 28 days before study enrollment until the end of the study

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
overall survival | three years
  compare to overall survival of patients who receive after 4 cycles of 5-azacytidine either allogeneic stem cell transplantation or continuous 5-azacytidine if no compatible donor is available overall 230 patients

SECONDARY OUTCOMES:
response | three years
  Comparison of response according to International Working Group Response Criteria between both arms:
  - Examinations of bone marrow (count of blasts) and peripheral blood (hematological improvement)after schedule of study assessments (after cycle 4 in both arms, after cycle 8 and after months 12-24-36 in the 5-azacytidine treatment and on day 100, day 180, months 12-24-36 after allogeneic stem cell transplantation
event-free survival | three years
  comparison of event free survival in both arms (230 pat.):
  - evaluation of survival status (relapse, date of relapse, alive or death) in the whole study period
overall survival | three years
  Comparison of overall survival between both arms (230 pat.).
  - evaluation of survival status (alive or death/date of death) in the whole study period
impact of Comorbidity-index on outcome | three years
  impact of comorbidity-index on outcome after study entry and prior to allogeneic stem cell transplantation (according definitions and weighted scores of comorbidities by Sorror et al):
  * physical examination
  * laboratory values(creatinine,Alt, AST, bilirubin, etc.)
  * apparative diagnostics (echo,lufu,ECG)
Treatment-related mortality | three years
  compare treatment related mortality in both arms (230 pat.):
  - death according to treatment in both arms
Evaluation of toxicity | three years
  the evaluation of toxicity will be performed according to the reporting guidelines as per NCI CTCAE in the whole study period:
  * adverse events grade 3 and 4
  * cytopenia grade 3 and 4 only be reported as AE which are judged by the investigator as clinically relevant
quality of life | three years
  Comparison of quality of life between both arms with the quality of life core questionnaire QLQ-C30 and the treatment specific high-dose chemotherapy module QLQ HD-C29 to assess the quality of life of cancer patient. The questionnaire has to be answered after the fourth cycle, 6 months, 1 year, 2 years and 3 years after both treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus Kroeger, Prof., Principal Investigator — University Medical Centre Hamburg-Eppendorf, Stem-Cell-Transplantation
Locations (16):
- Germany (16):
  - Charité Campus Benjamin Franklin, Berlin
  - Uniklinikum Bonn, Bonn
  - Universität zu Köln, Cologne
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt am Main
  - Universitätsklinikum Göttingen, Göttingen
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Mannheim, Mannheim
  - Klinikum rechts der Isar, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg, Nuremberg
  - Medizinische Universitätsklinik II, Tübingen
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kroger N, Sockel K, Wolschke C, Bethge W, Schlenk RF, Wolf D, Stadler M, Kobbe G, Wulf G, Bug G, Schafer-Eckart K, Scheid C, Nolte F, Kronke J, Stelljes M, Beelen D, Heinzelmann M, Haase D, Buchner H, Bleckert G, Giagounidis A, Platzbecker U. Comparison Between 5-Azacytidine Treatment and Allogeneic Stem-Cell Transplantation in Elderly Patients With Advanced MDS According to Donor Availability (VidazaAllo Study). J Clin Oncol. 2021 Oct 20;39(30):3318-3327. doi: 10.1200/JCO.20.02724. Epub 2021 Jul 20. PMID 34283629